CLINICAL TRIAL: NCT03419533
Title: An Observational Cross-sectional Study to Assess Oropharyngeal Carriage of N. Meningitidis in South Australian School Leavers
Brief Title: Study to Assess Oropharyngeal Carriage of N. Meningitidis in South Australian School Leavers
Acronym: B Part Of It
Status: Completed | Type: Observational
Sponsor: University of Adelaide (Other)
Responsible Party: Principal Investigator, Helen Marshall, Professor, University of Adelaide
Other Study IDs: HREC/16/WCHN/140_3
Record Dates: First submitted 2018-01-17; First posted 2018-02-05 (Actual); Results first posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Neisseria Meningitidis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Oropharyngeal throat swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 2018 school leavers: South Australian school leavers in 2018 (year 12 in 2017)
- 2019 school leavers: South Australian school leavers in 2019 (year 12 in 2018)

SUMMARY:
This is an observational cross sectional study to evaluate the impact of a 4CMenB vaccination program on oropharyngeal N. meningitidis carriage in vaccinated and unvaccinated school leavers.

DETAILED DESCRIPTION:
This carriage study of a cohort of school leavers in South Australia (SA) will provide an opportunity to assess carriage rates in the young adult population (school leavers) following introduction of a 4CMenB vaccination program in senior school students from 2017-2018.This will allow a comparison of carriage prevalence in the two years (2018 and 2019) following implementation of the school program to assess impact on carriage at a population level and compare carriage prevalence in vaccinated versus non-vaccinated groups. Assessment of any association between risk factors and prevalence of nasopharyngeal carriage in school leavers will be made and compared between vaccinated and unvaccinated students.

School leavers are defined as students who were enrolled in year 12 at school in the preceding year of recruitment and have been chosen as they are likely to have the highest carriage rates. A high proportion (approximately two thirds) of students will be immunised by the time of throat swab collection in years 2018 and 2019. Assessing carriage in both vaccinated and unvaccinated cohorts will further inform the effect of 4CMenB vaccine on carriage at a population level. This will help determine any herd immunity impact of 4CMenB vaccine and persistence of any effect.

ELIGIBILITY:
Inclusion Criteria:

* South Australian school leavers between 17 to 25 years of age (enrolled in year 12 in the previous year ie year 2018, students are eligible if they were enrolled in year 12 in 2017, year 2019, students are eligible if they were enrolled in year 12 in 2018).

Exclusion Criteria:

* No exclusion criteria

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: School leavers recruited through tertiary education sites and mail out through schools.
Sampling Method: Non-Probability Sample
Enrollment: 6802 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Marshall, Principal Investigator — University of Adelaide
Locations (1):
- Women's and Children's Hosptial, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Marshall HS, McMillan M, Koehler A, Lawrence A, MacLennan J, Maiden M, Ramsay M, Ladhani SN, Trotter C, Borrow R, Finn A, Sullivan T, Richmond P, Kahler C, Whelan J, Vadivelu K. B Part of It School Leaver protocol: an observational repeat cross-sectional study to assess the impact of a meningococcal serogroup B (4CMenB) vaccine programme on carriage of Neisseria meningitidis. BMJ Open. 2019 May 6;9(5):e027233. doi: 10.1136/bmjopen-2018-027233. PMID 31064808
- [Derived] McMillan M, Bednarz J, Leong LEX, Lawrence A, Marshall HS. Impact of COVID-19 Containment Strategies and Meningococcal Conjugate ACWY Vaccination on Meningococcal Carriage in Adolescents. Pediatr Infect Dis J. 2022 Nov 1;41(11):e468-e474. doi: 10.1097/INF.0000000000003660. Epub 2022 Jul 27. PMID 35895880
- [Derived] McMillan M, Koehler AP, Lawrence A, Sullivan TR, Bednarz J, MacLennan JM, Maiden MCJ, Ladhani SN, Ramsay ME, Trotter C, Borrow R, Finn A, Kahler CM, Whelan J, Vadivelu K, Richmond PC, Marshall HS. B Part of It School Leaver Study: A Repeat Cross-Sectional Study to Assess the Impact of Increasing Coverage With Meningococcal B (4CMenB) Vaccine on Carriage of Neisseria meningitidis. J Infect Dis. 2022 Feb 15;225(4):637-649. doi: 10.1093/infdis/jiab444. PMID 34487174

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 2018 School Leavers | 2019 School Leavers
Started | 4107 | 2695
Completed | 4107 | 2695
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2018 School Leavers | 2019 School Leavers | Total
Number analyzed (Participants) | 4107 | 2695 | 6802
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 18.45 (0.71) | 18.49 (0.51) | 18.47 (0.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female: Female | 2400 | 1660 | 4060
  Female: Male | 1707 | 1035 | 2742
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Aboriginal | 60 | 25 | 85
  Torres Strait Islander | 7 | 5 | 12
  Caucasian | 3063 | 1868 | 4931
  Asian | 440 | 467 | 907
  Middle Eastern | 66 | 58 | 124
  African | 66 | 49 | 115
  Pacific Islander | 6 | 11 | 17
  Other | 231 | 131 | 362
  Missing | 168 | 81 | 249

OUTCOME MEASURES:

1. Primary Outcome: Estimate the Difference in Carriage Prevalence of Disease Associated Genogroups of N. Meningitidis (A, B, C, W, X, Y) Between School Leavers in 2018 (Year 12 in 2017) and 2019 (Year 12 in 2018), Following a 4CMenB School Immunisation Program
Description: As measured by PCR in school leavers in 2018 and 2019
Time Frame: 2018 to 2019
Measure: Count of Participants; unit: Participants
Groups:
- 2018 School Leavers; 2019 School Leavers: Disease associated genogroups
Arm/Group | 2018 School Leavers | 2019 School Leavers
Number analyzed (Participants) | 4104 | 2690
Participants | 225 | 134

2. Secondary Outcome: Estimate the Difference in Carriage Prevalence of All N. Meningitidis Genogroups Between South Australian School Leavers in 2018 (Year 12 in 2017) and 2019 (Year 12 in 2018)
Description: As measured by PCR in school leavers in 2018 and 2019
Time Frame: 2018 to 2019
Measure: Count of Participants; unit: Participants
Groups:
- 2018 School Leavers; 2019 School Leavers: All genogroups
Arm/Group | 2018 School Leavers | 2019 School Leavers
Number analyzed (Participants) | 4104 | 2690
Participants | 393 | 227

3. Secondary Outcome: Estimate the Difference in Carriage Prevalence of Each N. Meningitidis Genogroup (A, B, C, W, X, Y) Between South Australian School Leavers in 2018 (Year 12 in 2017) and 2019 (Year 12 in 2018)
Description: As measured by PCR in school leavers in 2018 and 2019
Time Frame: 2018 to 2019
Measure: Count of Participants; unit: Participants
Groups:
- 2018 School Leavers; 2019 School Leavers: Each genogroup
Arm/Group | 2018 School Leavers | 2019 School Leavers
Number analyzed (Participants) | 4104 | 2690
Participants
  Group B | 86 | 64
  Group C | 16 | 8
  Group W | 21 | 4
  Group X | 1 | 6
  Group Y | 105 | 57
  Group E | 23 | 7
  Non groupable | 168 | 93

4. Secondary Outcome: Across Years, Estimate the Difference in Carriage Prevalence of N. Meningitidis Genogroups Causing Disease (A, B, C, W, X, Y) Between South Australian School Leavers Who Received 4CMenB Vaccine and Unvaccinated Students
Description: As measured by PCR in vaccinated and unvaccinated school leavers
Time Frame: 2018 to 2019
Measure: Count of Participants; unit: Participants
Groups:
- Vaccinated: 4CMenB vaccinated school leavers
- Unvaccinated: 4CMenB unvaccinated school leavers
Arm/Group | Vaccinated | Unvaccinated
Number analyzed (Participants) | 3885 | 2909
Participants | 200 | 159

5. Secondary Outcome: Across Years, Estimate the Difference in Carriage Prevalence of All N. Meningitidis Genogroups Between South Australian School Leavers Who Have Received 4CMenB and Unvaccinated Students.
Description: As measured by PCR in vaccinated and unvaccinated school leavers in 2018 and 2019
Time Frame: 2018 to 2019
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated | Unvaccinated
Number analyzed (Participants) | 3885 | 2909
Participants | 339 | 281

6. Secondary Outcome: Across Years, Estimate the Difference in Each N. Meningitidis Genogroup (A, B, C, W, X, Y) Carriage Prevalence Between South Australian School Leavers Who Received 4CMenB Vaccine and Unvaccinated Students
Description: As measured by PCR in vaccinated and unvaccinated school leavers
Time Frame: 2018 to 2019
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated | Unvaccinated
Number analyzed (Participants) | 3885 | 2909
Participants
  Group B | 83 | 67
  Group C | 11 | 13
  Group W | 9 | 16
  Group X | 6 | 1
  Group Y | 95 | 67
  Group E | 14 | 16
  Non-groupable | 139 | 122

7. Secondary Outcome: Identify Characteristics Associated With Carriage Prevalence of All N. Meningitidis Genogroups in South Australian School Leavers in 2018/2019
Description: As measured by PCR in school leavers
Time Frame: 2018 to 2019
Measure: Count of Participants; unit: Participants
Groups:
- Male; Female: Carriage prevalence of all N. meningitidis genogroups based on gender
Arm/Group | Male | Female
Number analyzed (Participants) | 2709 | 4055
Participants | 268 | 350

8. Secondary Outcome: Identify Characteristics Associated With Carriage Prevalence of N. Meningitidis Genogroups Causing Disease (A, B, C, W, X, Y) in South Australian School Leavers in 2018 /2019
Description: As measured by PCR in school leavers
Time Frame: 2018 to 2019
Measure: Count of Participants; unit: Participants
Arm/Group | Male | Female
Number analyzed (Participants) | 2709 | 4055
Participants | 154 | 204

9. Other Pre Specified Outcome: Describe Carriage Density of N. Meningitidis Genogroups as Measured by qPCR in School Leavers
Description: Density of N. meningitides by qPCR
Time Frame: 2018 to 2019
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Describe Genome Sequencing of Pathogenic N. Meningitidis (A, B, C, W, X, Y) in Carriage Among School Leavers.
Description: Whole genome sequencing of N. meningitidis
Time Frame: 2018 to 2019
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 years
Description: No adverse effects expected
Arm/Group | 2018 School Leavers | 2019 School Leavers
All-Cause Mortality (participants affected / at risk) | 0/4104 | 0/2690
Serious Adverse Events (participants affected / at risk) | 0/4104 | 0/2690
Other Adverse Events (participants affected / at risk) | 0/4104 | 0/2690

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-11-07): https://cdn.clinicaltrials.gov/large-docs/33/NCT03419533/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/33/NCT03419533/SAP_001.pdf